CLINICAL TRIAL: NCT00754650
Title: ML21206 - Bevacizumab in Chronic Lymphocytic Leukemia: A Proof of Concept Study
Brief Title: A Proof of Concept Study of the Safety, Tolerability, and Efficacy of Avastin (Bevacizumab) in Patients With Chemo-naive Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21206; 2007-004824-19 (EudraCT Number)
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Results first posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-05

CONDITIONS: Lymphocytic Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bevacizumab

ARMS (1):
- Bevacizumab 15 mg/kg (Experimental): Participants received bevacizumab 15 mg/kg intravenously on Day 1 of each 3-week cycle for 8 cycles.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab was supplied as a sterile liquid in single-use vials.
  Other Names: Avastin

SUMMARY:
This single arm study evaluated the bone marrow response, safety, and tolerability of 6 months treatment with Avastin (bevacizumab) monotherapy in patients with chronic lymphocytic leukemia. Patients received 8 cycles (21 days duration) of Avastin monotherapy (15mg/kg) with 6 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, ≥ 18 years of age.
* B-chronic lymphocytic leukemia not yet requiring treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* No previous treatment of chronic lymphocytic leukemia (CLL) by chemotherapy, radiotherapy, or immunotherapy.
* Life expectancy > 6 months.

Exclusion Criteria:

* Central nervous system (CNS) involvement by lymphoma or any evidence of spinal cord compression.
* Computed tomography (CT) scan based evidence of tumor invading major blood vessels.
* Gastrointestinal (GI) tract involvement by CLL.
* Active viral, bacterial, or fungal infection.
* Uncontrolled hypertension, cerebrovascular accident/stroke (≤ 6 months prior to randomization), myocardial infarction (≤ 6 months prior to randomization), unstable angina (≥ New York Heart Association (NYHA) Grade IV), thrombosis within 6 months before enrollment, NYHA Grade II congestive heart failure, or serious cardiac arrhythmia requiring ongoing medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Salzburg, Austria

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab 15 mg/kg
Started | 2
Completed | 0
Not Completed | 2
Not completed — Disease Progression | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All participants who received at least 1 administration of the study drug.
Arm/Group | Bevacizumab 15 mg/kg
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Bone Marrow Response
Description: Bone marrow response was defined as the change in percentage of infiltration at the interim staging (after 4 cycles of treatment) and the end of treatment.
Time Frame: Baseline to the end of treatment (up to 24 weeks)
Population: Intent-to-treat population: All participants who received at least 1 administration of the study drug.
Measure: Median (Inter-Quartile Range); unit: Percentage of infiltration
Arm/Group | Bevacizumab 15 mg/kg
Number analyzed (Participants) | 2
Percentage of infiltration
  Interim staging | -20.0 [-40.0 to 0.0]
  End of treatment | -20.0 [-40.0 to 0.0]

2. Secondary Outcome: Best Overall Response (BOR)
Description: The percentage of participants in each BOR category (complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD)) is reported. CR was defined as the disappearance of all target (TL) and non-target lesions (non-TL). PR was defined as ≥ 30% decrease in the sum of the longest diameter (SLD) of TLs, taking as reference the baseline SLD, or the persistence of 1 or more non-TLs. For TLs, SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest SLD since treatment started. For non-TLs, SD was defined as the persistence of 1 or more lesions. PD was defined as ≥ 20% increase in the sum of the longest diameter of TLs, taking as reference the smallest SLD recorded since treatment started, the unequivocal progression of existing non-TLs, or the appearance of 1 or more new lesions.
Time Frame: Baseline to the end of treatment (up to 24 weeks)
Population: Intent-to-treat population: All participants who received at least 1 administration of the study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab 15 mg/kg
Number analyzed (Participants) | 2
Percentage of participants
  Interim staging - Complete response | 0.0
  Interim staging - Partial response | 0.0
  Interim staging - Stable disease | 50.0
  Interim staging - Progressive disease | 50.0
  End of treatment - Complete response | 0.0
  End of treatment - Partial response | 0.0
  End of treatment - Stable disease | 0.0
  End of treatment - Progressive disease | 100.0

ADVERSE EVENTS:
Description: Intent-to-treat population: All participants who received at least 1 administration of the study drug.
Arm/Group | Bevacizumab 15 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab 15 mg/kg (N=2)
Nasopharyngitis (Infections and infestations) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.